CLINICAL TRIAL: NCT05555290
Title: ALTA - ALbuterol/Budesonide Treatment in Acute Airway Obstruction. A Randomized, Double-blind, 2-period, Cross-over Study Evaluating Efficacy and Safety of Repeated Doses of PT027 Compared to PT007 in Patients With Asthma and Acute Airway Obstruction Induced by Repeated Mannitol Challenges
Brief Title: PT027 Compared to PT007 in Patients With Asthma With Mannitol-induced Acute Airway Obstruction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6930C00017
Record Dates: First submitted 2022-08-25; First posted 2022-09-26 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Asthma
Keywords: Acute airway obstruction; Albuterol; Budesonide; Short-acting beta2-agonists (SABA); Albuterol Sulfate
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: The study will enroll 17 participants in Part 1 and 88 participants in Part 2
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (PT027) [experimental], then Treatment B (PT007) [active comparator] Part 1 & 2 (Experimental): At Visit 2, participants will receive repeated oral inhalations of PT027 to treat acute airway obstruction induced by a repeated airway challenge, followed by a washout period of 10-14 days. At Visit 3, participants will receive repeated oral inhalations of PT007 to treat acute airway obstruction induced by a repeated airway challenge.
  Interventions: Combination Product: PT027; Combination Product: PT007
- Treatment B (PT007) [active comparator], then Treatment A (PT027) [experimental] Part 1 & 2 (Experimental): At Visit 2, participants will receive repeated oral inhalations of PT007 to treat acute airway obstruction induced by a repeated airway challenge, followed by a washout period of 10 to 14 days. At Visit 3, participants will receive repeated oral inhalations of PT027 to treat acute airway obstruction induced by a repeated airway challenge.
  Interventions: Combination Product: PT027; Combination Product: PT007

INTERVENTIONS:
Combination Product: PT027 — When administered PT027, participants will receive 2 actuations of albuterol- budesonide per dose administered as oral inhalations.
Combination Product: PT007 — When administered PT007, participants will receive 2 actuations of albuterol administered as oral inhalations.

SUMMARY:
A study evaluating efficacy and safety of repeated doses of PT027 compared to PT007 in patients with asthma and acute airway obstruction induced by repeated mannitol challenges

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, 2-period, cross-over study evaluating efficacy and safety of repeated doses of PT027 (albuterol/budesonide pressurized metered dose inhaler (pMDI)) compared to PT007 (albuterol pMDI) in participants with asthma and acute airway obstruction induced by 2 mannitol challenges at least 8 hours apart.

It is a two-part study where Part 1 will enroll a small cohort of participants and will be used as a pilot study. The data obtained from Part 1 will be assessed by an internal AstraZeneca advisory board, and suggested changes may be made to Part 2 of the study.

The following is the sequence of study visits:

(i) Visit 1 (V1) screening (ii) Visit 2 (V2) 10 to 14 days after Visit 1 assessments; 1st dual challenge and treatment visit (iii) Visit 3 (V3) 10 to 14 days after Visit 2; 2nd dual challenge and treatment visit

At Visit 1, all participants will be subjected to a single mannitol challenge to establish a positive response (defined as a ≥15% decrease in forced expiratory volume in the first second [FEV1] from the 0 mg mannitol FEV1 value) and will receive 4 puffs of open-label PT007. At Visit 2, participants will be randomized to one of 2 treatment sequences, A/B or B/A, where treatments A and B are defined as:

(i) Treatment A = PT027 (ii) Treatment B = PT007

For treatment sequence A/B, participants will receive repeated inhalations of PT027 at Visit 2 followed by repeated inhalations of PT007 in Visit 3 .

For treatment sequence B/A, participants will receive repeated inhalations of PT007 at Visit 2 followed by repeated inhalations of PT027 in Visit 3.

Participants will have a Follow-up Telephone call 7 days after Visit 3/after Early discontinuation (ED).

ELIGIBILITY:
Inclusion Criteria:

* Participants who have been diagnosed with asthma > 6 months before Visit 1 by a physician.
* Participants must have been prescribed and using as-needed SABA as only asthma treatment for at least 4 weeks before screening visit.
* Participants should have pre-bronchodilator FEV1 ≥ 1.5 L and FEV1 ≥ 60% to < 90% predicted normal at Visit 1.
* Participants should have a positive response to mannitol challenge performed at Visit 1 (a decrease in FEV1 by at least 15% [PD15] at ≤ 635 mg).
* Participants should return to within 10% of baseline FEV1 (≥ 90% of baseline FEV1), within 1 hour after positive mannitol challenge and 4 inhalations of PT007, performed at Visit 1.
* Participants should be able to adhere to study procedures in the judgment of the Investigator.
* Male or female.
* Women of childbearing potential must have a negative urine pregnancy test at each study visit.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and in this protocol.
* Provision of signed and dated written Optional Genetic Research Information informed consent prior to collection of samples for optional genetic research that supports Genomic Initiative.

Exclusion Criteria:

* Any evidence of clinically significant lung disease other than asthma.
* If the participant has had any face-to-face unscheduled or urgent visit for asthma worsening within the last 4 weeks.
* Any significant disease or disorder, or evidence of drug/substance abuse which in the Investigator's opinion would pose a risk to participant safety, interfere with the conduct of study, have an impact on the study results, or make it undesirable for the participant to participate in the study.
* If participants have used Inhaled corticosteroids (ICS) within 1 month prior to enrolment.
* If they have used immunosuppressive medication (including but not limited to methotrexate, troleandomycin, cyclosporine, azathioprine, systemic corticosteroids including regular treatment with oral corticosteroids or intramuscular long-acting depot corticosteroids, or any experimental anti-inflammatory therapy) within 3 months prior to enrolment (Visit 1) or plan on starting immunosuppressive medications during the study.
* If they have used allergen-specific immunotherapy (desensitization) within 3 months prior to enrolment.
* If they have used systemic corticosteroids (including oral and injected) within 3 months prior to enrolment.
* If they have received any marketed or investigational biologic within 4 months or 5 half-lives prior to enrolment (whichever is longer) or received any investigational nonbiologic agent within 30 days or 5 half-lives prior to enrolment (whichever is longer).
* Participants with a known hypersensitivity to beta2-agonists, ICS, mannitol, or any of the excipients of the product.
* Any clinically significant abnormal findings in physical examination, vital signs, ECG (eg, participants with QTcF > 500 ms), hematology, clinical chemistry, or urinalysis, which in the opinion of the Investigator, may put the participant at risk because of his/her participation in the study, or may influence the results of the study, or the participant's ability to complete entire duration of the study.
* If they are current smokers or participants with smoking history ≥ 10 pack years including the use of vaping products, such as electronic cigarettes, and water pipes. If they are former smokers with a smoking history of <10 pack years, including former vaping or water pipe users, smoking must have stopped for at least 6 months prior to Visit 1 to be eligible.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and its affiliates and/or staff at the study site and their immediate relative(s)).
* Judgment by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
* Breast feeding, pregnancy or intention to become pregnant during the course of the study.
* Previous randomization in the present study.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Columbia, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6930C00017&attachmentIdentifier=5d689e8b-41b8-4e67-bdd0-1ea82e0a1c08&fileName=AZ_EMPOWER_D6930C00017_ALTA_(PXL_264369)_CSR_Synopsis_no_redaction_Final_PDF-A.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 28 September 2022 to 18 November 2024 at 11 study centers in the United States of America (USA).
  Participants were enrolled separately to Part 1 and Part 2 of the study. Both parts were conducted independently and no cross-over happened between the parts.
Pre-assignment Details: Participants who signed informed consent form (ICF) were enrolled into the study and those who met all eligibility criteria during screening were randomized and treated. All study assessments were performed as per the schedule.
  A total of 190 participants who provided the ICF were enrolled and screened at Visit 1. Of these, 105 participants met the eligibility criteria at Visit 2 and were randomized and treated in the study; thus, only data for these participants was collectable and analyzable.
Groups:
- Treatment A (PT027) [Experimental], Then Treatment B (PT007) [Active Comparator] Part 1 & 2: At Visit 2, participants received repeated oral inhalations of PT027 to treat acute airway obstruction induced by a repeated airway challenge, followed by a washout period of 10-14 days. At Visit 3, participants received repeated oral inhalations of PT007 to treat acute airway obstruction induced by a repeated airway challenge.
- Treatment B (PT007) [Active Comparator], Then Treatment A (PT027) [Experimental] Part 1 & 2: At Visit 2, participants received repeated oral inhalations of PT007 to treat acute airway obstruction induced by a repeated airway challenge, followed by a washout period of 10 to 14 days. At Visit 3, participants received repeated oral inhalations of PT027 to treat acute airway obstruction induced by a repeated airway challenge.
Period: Part 1
Arm/Group | Treatment A (PT027) [Experimental], Then Treatment B (PT007) [Active Comparator] Part 1 & 2 | Treatment B (PT007) [Active Comparator], Then Treatment A (PT027) [Experimental] Part 1 & 2
Started | 8 | 9
Completed | 7 | 8
Not Completed | 1 | 1
Not completed — Development of study-specific withdrawal criteria | 1 | 1
Period: Part 2
Arm/Group | Treatment A (PT027) [Experimental], Then Treatment B (PT007) [Active Comparator] Part 1 & 2 | Treatment B (PT007) [Active Comparator], Then Treatment A (PT027) [Experimental] Part 1 & 2
Started | 44 | 44
Completed | 41 | 40
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Early termination | 0 | 3

BASELINE CHARACTERISTICS:
Population: All participants randomly assigned to any of the 2 study treatment sequences and who took at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A (PT027) [Experimental], Then Treatment B (PT007) [Active Comparator] Part 1 & 2 | Treatment B (PT007) [Active Comparator], Then Treatment A (PT027) [Experimental] Part 1 & 2 | Total
Number analyzed (Participants) | 52 | 53 | 105
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.1 (13.1) | 43.3 (13.3) | 44.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 25 | 62
  Male | 15 | 28 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 8 | 20
  Not Hispanic or Latino | 40 | 45 | 85
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Change From Mannitol Baseline Forced Expiratory Volume in the First Second (FEV1) Area Under the Curve (AUC [0-60 Min]) Post-mannitol Challenge 1 - Non-Inferiority Analysis
Description: The efficacy of repeated dosing of PT027 relative to PT007, on post-dose lung function, when used by participants with asthma on SABA as-needed treatment only who are experiencing acute airway obstruction induced by mannitol challenges was assessed.
  Mannitol baseline was defined as the FEV1 result where a positive response to mannitol was observed prior to dosing of study drug for challenge 1 in Visit 2 and in Visit 3 (time 0). A positive response was defined as a ≥ 15% decrease from the FEV1 determined after the 0 mg mannitol dose up to ≤ 635 mg cumulative mannitol dose.
  The primary efficacy comparison of non-inferiority of PT027 versus PT007 evaluated the while-on treatment estimand in the Per Protocol (PP) analysis set and was based on a 1-sided hypothesis testing approach with a non-inferiority margin of -150 mL.
Time Frame: Up to 60 minutes post mannitol challenge 1
Population: PP analysis set included all participants who received all doses of study treatment following mannitol challenge 1, had baseline and post-treatment study evaluation (spirometry tests), and did not have any important protocol deviations. Challenge 1 referred to the first mannitol challenge for Visits 2 and 3.
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Groups:
- Treatment A (PT027) [Experimental]: Participants received repeated oral inhalations (2 actuations) of PT027 to treat acute airway obstruction induced by a repeated airway challenge.
- Treatment B (PT007) [Active Comparator]: Participants received repeated oral inhalations (2 actuations) of PT007 to treat acute airway obstruction induced by a repeated airway challenge.
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 15 | 15
milliliters (mL) | 638.7 (206.4) | 657.9 (284.4)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Non-Inferiority — Non-inferiority was established if the lower 95% confidence limit of the point estimate of the treatment effect was greater than the non-inferiority margin of -150 mL; Difference in least squares means = -6.24, 95% CI 2-sided [-60.52 to 48.04] — The analysis was performed using a linear mixed effects model. The dependent variable was change from mannitol baseline in AUC0-60 min (in mL) post mannitol challenge 1

2. Primary Outcome: Part 1: Change From Mannitol Baseline FEV1 AUC (0-60 Min) Post-mannitol Challenge 1 - Superiority Analysis
Description: The efficacy of repeated dosing of PT027 relative to PT007, on post-dose lung function, when used by participants with asthma on SABA as-needed treatment only who are experiencing acute airway obstruction induced by mannitol challenges was assessed.
  Mannitol baseline was defined as the FEV1 result where a positive response to mannitol was observed prior to dosing of study drug for challenge 1 in Visit 2 and in Visit 3 (time 0). A positive response was defined as a ≥ 15% decrease from the FEV1 determined after the 0 mg mannitol dose up to ≤ 635 mg cumulative mannitol dose.
  If non-inferiority was demonstrated, then comparisons were made to establish the superiority of PT027 versus PT007. The primary efficacy comparison of superiority was based on a 2-sided hypothesis testing approach in the randomized set (RS). Superiority was concluded if the 2-sided p-value was < 0.05.
Time Frame: Up to 60 minutes post mannitol challenge 1
Population: RS included all participants who were randomized to any of the 2 treatment sequences, A/B or B/A.
  Treatments A and B were defined as:
  Treatment A = PT027 180/160 µg pressurized metered dose inhaler (pMDI) Treatment B = PT007 180 µg pMDI
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 16 | 15
milliliters (mL) | 624.2 (207.6) | 657.9 (284.4)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Superiority; p = 0.762, Linear mixed effects model; Difference in least squares means = -7.71, 95% CI 2-sided [-61.95 to 46.54] — The analysis was performed using a linear mixed-effects model. The dependent variable was the change from mannitol baseline in AUC(0-60 min) (in mL) post-mannitol challenge 1

3. Primary Outcome: Part 2: Change From Mannitol Baseline FEV1 AUC (0-60 Min) Post-mannitol Challenge 1 - Non-Inferiority Analysis
Description: The efficacy of repeated dosing of PT027 relative to PT007, on post-dose lung function, when used by participants with asthma on SABA as-needed treatment only who are experiencing acute airway obstruction induced by mannitol challenges was assessed.
  Mannitol baseline was defined as the FEV1 result where a positive response to mannitol was observed prior to dosing of study drug for challenge 1 in Visit 2 and in Visit 3 (time 0). A positive response was defined as a ≥ 15% decrease from the FEV1 determined after the 0 mg mannitol dose up to ≤ 635 mg cumulative mannitol dose.
  The primary efficacy comparison of non-inferiority of PT027 versus PT007 evaluated the while-on-treatment estimand in the PP analysis set and was based on a 1-sided hypothesis testing approach with a non-inferiority margin of -150 mL.
Time Frame: Up to 60 minutes post mannitol challenge 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 67 | 67
milliliters (mL) | 749.7 (347.0) | 758.1 (342.3)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in least squares means = -9.14, 95% CI 2-sided [-55.53 to 37.25] — [estimate comment as in outcome 2, analysis 1]

4. Primary Outcome: Part 2: Change From Mannitol Baseline FEV1 AUC (0-60 Min) Post-mannitol Challenge 1 - Superiority Analysis
Description: The efficacy of repeated dosing of PT027 relative to PT007, on post-dose lung function, when used by participants with asthma on SABA as-needed treatment only who are experiencing acute airway obstruction induced by mannitol challenges was assessed.
  Mannitol baseline was defined as the FEV1 result where a positive response to mannitol was observed prior to dosing of study drug for challenge 1 in Visit 2 and in Visit 3 (time 0). A positive response was defined as a ≥ 15% decrease from the FEV1 determined after the 0 mg mannitol dose up to ≤ 635 mg cumulative mannitol dose.
  If non-inferiority was demonstrated, then comparisons were made to establish the superiority of PT027 versus PT007. The primary efficacy comparison of superiority was based on a 2-sided hypothesis testing approach in the modified randomized set (mRS). Superiority was concluded if the 2-sided p-value was < 0.05.
Time Frame: Up to 60 minutes post mannitol challenge 1
Population: mRS included all participants who were randomized to any of the 2 treatment sequences, A/B or B/A and received any amount of randomized study treatment.
  Treatments A and B were defined as:
  Treatment A = PT027 180/160 µg pMDI Treatment B = PT007 180 µg pMDI
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 84 | 85
milliliters (mL) | 688.6 (342.3) | 716.9 (348.3)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Superiority; p = 0.257, Linear mixed effects model; Difference in least squares means = -25.78, 95% CI 2-sided [-70.77 to 19.20] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Part 1: Change From Mannitol Baseline in FEV1 AUC (0-15 Min) Post-mannitol Challenge 1 - Non-Inferiority Analysis
Description: The efficacy of PT027 after a single dose compared with PT007 in reversal of acute airway obstruction, when used by participants with asthma on SABA as-needed treatment only who are experiencing acute airway obstruction induced by mannitol challenges was assessed.
  Mannitol baseline was defined as the FEV1 result where a positive response to mannitol was observed prior to dosing of study drug for challenge 1 in Visit 2 and in Visit 3 (time 0). A positive response was defined as a ≥ 15% decrease from the FEV1 determined after the 0 mg mannitol dose up to ≤ 635 mg cumulative mannitol dose.
  The efficacy comparison of non-inferiority of PT027 versus PT007 evaluated the while-on-treatment estimand in the PP analysis set and was based on a 1-sided hypothesis testing approach with a non-inferiority margin of -150 mL.
Time Frame: Up to 15 minutes post mannitol challenge 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 15 | 15
milliliters (mL) | 372.3 (156.9) | 391.4 (235.7)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in least squares means = -12.26, 95% CI 2-sided [-77.99 to 53.48] — The analysis was performed using a linear mixed-effects model. The dependent variable was change from mannitol baseline in AUC(0-15 min) (in mL) post-mannitol challenge 1

6. Secondary Outcome: Part 1: Change From Mannitol Baseline in FEV1 AUC (0-15 Min) Post-mannitol Challenge 1 - Superiority Analysis
Description: The efficacy of PT027 after a single dose compared with PT007 in reversal of acute airway obstruction, when used by participants with asthma on SABA as-needed treatment only who are experiencing acute airway obstruction induced by mannitol challenges was assessed.
  Mannitol baseline was defined as the FEV1 result where a positive response to mannitol was observed prior to dosing of study drug for challenge 1 in Visit 2 and in Visit 3 (time 0). A positive response was defined as a ≥ 15% decrease from the FEV1 determined after the 0 mg mannitol dose up to ≤ 635 mg cumulative mannitol dose.
  If non-inferiority was demonstrated, then comparisons were made to establish the superiority of PT027 versus PT007. The primary efficacy comparison of superiority was based on a 2-sided hypothesis testing approach in the RS. Superiority was concluded if the 2-sided p-value was < 0.05.
Time Frame: Up to 15 minutes post mannitol challenge 1
Population: RS included all participants who were randomized to any of the 2 treatment sequences, A/B or B/A.
  Treatments A and B were defined as:
  Treatment A = PT027 180/160 µg pMDI Treatment B = PT007 180 µg pMDI
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Groups:
- Treatment A (PT027) [Experimental]: Participants received repeated oral inhalations of PT027 (2 actuations) to treat acute airway obstruction induced by a repeated airway challenge.
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 16 | 15
milliliters (mL) | 367.4 (152.8) | 391.4 (235.7)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Superiority; p = 0.656, Linear mixed effects model; Difference in least squares means = -13.69, 95% CI 2-sided [-79.05 to 51.66] — The analysis was performed using a linear mixed-effects model. The dependent variable was the change from mannitol baseline in AUC0-15 min (in mL) post-mannitol challenge 1

7. Secondary Outcome: Part 2: Change From Mannitol Baseline in FEV1 AUC (0-15 Min) Post-mannitol Challenge 1 - Non-Inferiority Analysis
Description: as for outcome 5
Time Frame: Up to 15 minutes post mannitol challenge 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 67 | 67
milliliters (mL) | 476.6 (267.8) | 496.4 (267.6)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in least squares means = -20.46, 95% CI 2-sided [-71.13 to 30.21] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Part 2: Change From Mannitol Baseline in FEV1 AUC (0-15 Min) Post-mannitol Challenge 1 - Superiority Analysis
Description: The efficacy of PT027 after a single dose compared with PT007 in reversal of acute airway obstruction, when used by participants with asthma on SABA as-needed treatment only who are experiencing acute airway obstruction induced by mannitol challenges was assessed.
  Mannitol baseline was defined as the FEV1 result where a positive response to mannitol was observed prior to dosing of study drug for challenge 1 in Visit 2 and in Visit 3 (time 0). A positive response was defined as a ≥ 15% decrease from the FEV1 determined after the 0 mg mannitol dose up to ≤ 635 mg cumulative mannitol dose.
  If non-inferiority was demonstrated, then comparisons were made to establish the superiority of PT027 versus PT007. The primary efficacy comparison of superiority was based on a 2-sided hypothesis testing approach in the mRS. Superiority was concluded if the 2-sided p-value was < 0.05.
Time Frame: Up to 15 minutes post mannitol challenge 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 84 | 85
milliliters (mL) | 435.8 (260.3) | 469.8 (272.2)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Superiority; p = 0.195, Linear mixed effects model; Difference in least squares means = -31.56, 95% CI 2-sided [-79.60 to 16.47] — The analysis was performed using a linear mixed-effects model. The dependent variable was the change from mannitol baseline in AUC(0-15 min) (in mL) post-mannitol challenge 1

9. Secondary Outcome: Part 1: Change From Mannitol Baseline in FEV1 at 7 Hours Post-mannitol Challenge 1 - Non-Inferiority Analysis
Description: The efficacy of PT027 compared with PT007 in the sustainability of effect of reversal of acute airway obstruction post-mannitol challenge 1 in participants with asthma on SABA as needed treatment only who are experiencing acute airway obstruction induced by mannitol challenges was assessed.
  Mannitol baseline was defined as the FEV1 result where a positive response to mannitol is observed prior to dosing of study drug for challenge 1 in Visit 2 and in Visit 3 (time 0). A positive response was defined as a ≥ 15% decrease from the FEV1 determined after the 0 mg mannitol dose up to ≤ 635 mg cumulative mannitol dose.
  The efficacy comparison of non-inferiority of PT027 versus PT007 evaluated the while-on-treatment estimand in the PP analysis set and was based on a 1-sided hypothesis testing approach with a non-inferiority margin of -150 mL.
Time Frame: At 7 hours post mannitol challenge 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 15 | 15
milliliters (mL) | 680.7 (207.1) | 728.6 (274.3)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in least squares means = -32.96, 95% CI 2-sided [-106.29 to 40.37] — The analysis was performed using a linear mixed-effects model. The dependent variable was change from mannitol baseline in FEV1 result (in mL) at 7 hours post mannitol challenge 1

10. Secondary Outcome: Part 1: Change From Mannitol Baseline in FEV1 at 7 Hours Post-mannitol Challenge 1 - Superiority Analysis
Description: The efficacy of PT027 compared with PT007 in the sustainability of effect of reversal of acute airway obstruction post-mannitol challenge 1 in participants with asthma on SABA as needed treatment only who are experiencing acute airway obstruction induced by mannitol challenges was assessed.
  Mannitol baseline was defined as the FEV1 result where a positive response to mannitol was observed prior to dosing of study drug for challenge 1 in Visit 2 and in Visit 3 (time 0). A positive response was defined as a ≥ 15% decrease from the FEV1 determined after the 0 mg mannitol dose up to ≤ 635 mg cumulative mannitol dose.
  If non-inferiority was demonstrated, then comparisons were made to establish the superiority of PT027 versus PT007. The primary efficacy comparison of superiority was based on a 2-sided hypothesis testing approach in the RS. Superiority was concluded if the 2-sided p-value was < 0.05.
Time Frame: At 7 hours post mannitol challenge 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 16 | 15
milliliters (mL) | 662.2 (213.4) | 728.6 (274.3)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Superiority; p = 0.303, Linear mixed effects model; Difference in least squares means = -36.29, 95% CI 2-sided [-109.71 to 37.13] — The analysis was performed using a linear mixed-effects model. The dependent variable was the change from mannitol baseline in FEV1 result (in mL) at 7 hours post-mannitol challenge 1

11. Secondary Outcome: Part 2: Change From Mannitol Baseline in FEV1 at 480 Minutes Post-mannitol Challenge 1 - Non-Inferiority Analysis
Description: The efficacy of PT027 compared with PT007 in the sustainability of effect of reversal of acute airway obstruction post-mannitol challenge 1 in participants with asthma on SABA as needed treatment only who are experiencing acute airway obstruction induced by mannitol challenges was assessed.
  Mannitol baseline was defined as the FEV1 result where a positive response to mannitol was observed prior to dosing of study drug for challenge 1 in Visit 2 and in Visit 3 (time 0). A positive response was defined as a ≥ 15% decrease from the FEV1 determined after the 0 mg mannitol dose up to ≤ 635 mg cumulative mannitol dose.
  The efficacy comparison of non-inferiority of PT027 versus PT007 evaluated the while-on-treatment estimand in the PP analysis set and was based on a 1-sided hypothesis testing approach with a non-inferiority margin of -150 mL.
Time Frame: At 480 minutes post mannitol challenge 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 66 | 67
milliliters (mL) | 765.8 (411.8) | 683.5 (375.2)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in least squares means = 91.09, 95% CI 2-sided [28.16 to 154.03] — The analysis was performed using a linear mixed-effects model. The dependent variable was the change from mannitol baseline in FEV1 result (in mL) at 480 min post-mannitol challenge 1

12. Secondary Outcome: Part 2: Change From Mannitol Baseline in FEV1 at 480 Minutes Post-mannitol Challenge 1 - Superiority Analysis
Description: The efficacy of PT027 compared with PT007 in the sustainability of effect of reversal of acute airway obstruction post-mannitol challenge 1 in participants with asthma on SABA as needed treatment only who are experiencing acute airway obstruction induced by mannitol challenges was assessed.
  Mannitol baseline was defined as the FEV1 result where a positive response to mannitol was observed prior to dosing of study drug for challenge 1 in Visit 2 and in Visit 3 (time 0). A positive response was defined as a ≥ 15% decrease from the FEV1 determined after the 0 mg mannitol dose up to ≤ 635 mg cumulative mannitol dose.
  If non-inferiority was demonstrated, then comparisons were made to establish the superiority of PT027 versus PT007. The primary efficacy comparison of superiority was based on a 2-sided hypothesis testing approach in the mRS. Superiority was concluded if the 2-sided p-value was < 0.05.
Time Frame: At 480 minutes post mannitol challenge 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 82 | 85
milliliters (mL) | 759.9 (395.1) | 684.5 (378.3)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Superiority; p = 0.001, Linear mixed effects model; Difference in least squares means = 91.19, 95% CI 2-sided [36.69 to 145.68] — The analysis is performed using a linear mixed-effects model. The dependent variable is change from mannitol baseline in FEV1 result (in mL) at 480 min post-mannitol challenge 1

13. Secondary Outcome: Part 1: Time to Return to Baseline (-30 Min) FEV1 Post-mannitol Challenge 2 - Non-Inferiority Analysis
Description: The efficacy of a single dose of PT027 compared with PT007 on post-dose speed of recovery of lung function following a recurring trigger of acute airway obstruction induced by mannitol challenges in participants with asthma on SABA as needed treatment only was assessed.
  The time to return in minutes was calculated as the time it took for a participant to return to within 5% of the baseline (- 30 min) FEV1 value, post-mannitol challenge 2.
  FEV1 baseline is defined as the best FEV1 value (the highest FEV1 of the acceptable efforts) taken pre-mannitol challenge at - 30 min for Visit 2 and Visit 3.
  The efficacy comparison of non-inferiority of PT027 versus PT007 evaluated the while-on-treatment estimand in the PP analysis set and was based on a 1-sided hypothesis testing approach with a non-inferiority margin of 3.5 min.
Time Frame: From baseline (30 minutes prior to mannitol challenge 1) up to 60 minutes post-mannitol challenge 2 (up to 550 minutes post-mannitol challenge 1)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: minutes (min)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 15 | 15
minutes (min) | 8.5 [7.00 to 11.00] | 8.0 [6.00 to 15.00]
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Non-Inferiority — Non-inferiority was established if the upper 95% confidence limit of the point estimate of the treatment effect was less than the non-inferiority margin of 3.5 min; Median Difference (Final Values) = 0.50, 95% CI 2-sided [-1.50 to 2.00] — The analysis was performed using a Wilcoxon Signed-Rank Test

14. Secondary Outcome: Part 1: Time to Return to Baseline (-30 Min) FEV1 Post-mannitol Challenge 2 - Superiority Analysis
Description: The efficacy of a single dose of PT027 compared with PT007 on post-dose speed of recovery of lung function following a recurring trigger of acute airway obstruction induced by mannitol challenges in participants with asthma on SABA as needed treatment only was assessed.
  The time to return in minutes was calculated as the time it took for a participant to return to within 5% of the baseline (- 30 min) FEV1 value, post-mannitol challenge 2.
  FEV1 baseline was defined as the best FEV1 value (the highest FEV1 of the acceptable efforts) taken pre-mannitol challenge at - 30 min for Visit 2 and Visit 3.
  If non-inferiority was demonstrated, then comparisons were made to establish the superiority of PT027 versus PT007. The primary efficacy comparison of superiority was based on a 2-sided hypothesis testing approach in the RS. Superiority was concluded if the 2-sided p-value was < 0.05.
Time Frame: as for outcome 13
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: minutes (min)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 15 | 15
minutes (min) | 8.5 [7.00 to 11.00] | 8.0 [6.00 to 15.00]
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Superiority; p = 0.514, Wilcoxon Signed-Rank test; Median Difference (Final Values) = 0.50, 95% CI 2-sided [-1.50 to 2.00] — The analysis was performed using a Wilcoxon Signed-Rank Test

15. Secondary Outcome: Part 2: Time to Return to Baseline (-30 Min) FEV1 Post-mannitol Challenge 2, Pre-final Dose of Rescue/Reliever - Non-Inferiority Analysis
Description: The efficacy of a single dose of PT027 compared with PT007 on post-dose speed of recovery of lung function following a recurring trigger of acute airway obstruction induced by mannitol challenges in participants with asthma on SABA as needed treatment only was assessed.
  The time to return in minutes was calculated as the time it took for a participant to return to within 5% of the baseline (- 30 min) FEV1 value, post-mannitol challenge 2.
  FEV1 baseline was defined as the best FEV1 value (the highest FEV1 of the acceptable efforts) taken pre-mannitol challenge at - 30 min for Visit 2 and Visit 3.
  The efficacy comparison of non-inferiority of PT027 versus PT007 evaluated the while-on-treatment estimand in the modified per protocol (mPP) analysis set and was based on a 1-sided hypothesis testing approach with a non-inferiority margin of 3.5 min.
Time Frame: as for outcome 13
Population: mPP analysis set included all participants who received all doses of study treatment following mannitol challenge 1, had baseline and post-treatment study evaluation (spirometry tests) and did not have any important protocol deviations, apart from the deviation of not receiving first dose of investigational medical product (IMP) within 6 minutes of final dose of mannitol challenge 1 (IP03b). Challenge 1 referred to the first mannitol challenge for Visits 2 and 3.
Measure: Median (Inter-Quartile Range); unit: minutes (min)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 78 | 74
minutes (min) | 4.5 [4.0 to 7.0] | 4.0 [3.0 to 5.0]
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; Median Difference (Final Values) = 0.00, 95% CI 2-sided [-1.50 to 2.00] — The analysis was performed using a Wilcoxon Signed-Rank Test

16. Secondary Outcome: Part 2: Time to Return to Baseline (-30 Min) FEV1 Post-mannitol Challenge 2, Pre-final Dose of Rescue/Reliever - Superiority Analysis
Description: The efficacy of a single dose of PT027 compared with PT007 on post-dose speed of recovery of lung function following a recurring trigger of acute airway obstruction induced by mannitol challenges in participants with asthma on SABA as needed treatment only was assessed.
  The time to return in minutes was calculated as the time it took for a participant to return to within 5% of the baseline (- 30 min) FEV1 value, post-mannitol challenge 2.
  FEV1 baseline was defined as the best FEV1 value (the highest FEV1 of the acceptable efforts) taken pre-mannitol challenge at - 30 min for Visit 2 and Visit 3.
  If non-inferiority was demonstrated, then comparisons were made to establish the superiority of PT027 versus PT007. The primary efficacy comparison of superiority was based on a 2-sided hypothesis testing approach in the mRS. Superiority was concluded if the 2-sided p-value was < 0.05.
Time Frame: as for outcome 13
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: minutes (min)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 82 | 79
minutes (min) | 4.5 [4.0 to 7.0] | 4.0 [3.0 to 6.0]
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Superiority; p = 0.627, Wilcoxon Signed-Rank test; Median Difference (Final Values) = 0.50, 95% CI 2-sided [-1.50 to 2.00] — The analysis was performed using a Wilcoxon Signed-Rank Test

17. Secondary Outcome: Part 1: Peak Fall in FEV1 From Baseline (-30 Min) FEV1 to Post-mannitol Challenge 2, Pre-dose - Non-Inferiority Analysis
Description: The protective efficacy of prior repetitive doses of PT027 compared with PT007 on lung function fall in response to a recurring trigger of acute airway obstruction induced by mannitol challenges in participants with asthma on SABA as-needed treatment only was assessed.
  FEV1 baseline was defined as the best FEV1 value (the highest FEV1 of the acceptable efforts) taken pre-mannitol challenge at - 30 min for Visit 2 and Visit 3.
  FEV1 at post-mannitol challenge 2 was the FEV1 result recorded at the end of mannitol challenge 2, i.e. before study intervention treatment, was expected to be at ~490 mins following the mannitol challenge 1.
  The efficacy comparison of non-inferiority of PT027 versus PT007 evaluated the while-on-treatment estimand in the mPP analysis set and was based on a 1-sided hypothesis testing approach with a non-inferiority margin of -150 mL.
Time Frame: Baseline (30 minutes prior to mannitol challenge 1) and at 490 minutes post-mannitol challenge 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 15 | 15
milliliters (mL) | 87.1 (323.2) | 137.7 (302.9)

18. Secondary Outcome: Part 1: Peak Fall in FEV1 From Baseline (-30 Min) FEV1 to Post-mannitol Challenge 2, Pre-dose - Superiority Analysis
Description: The protective efficacy of prior repetitive doses of PT027 compared with PT007 on lung function fall in response to a recurring trigger of acute airway obstruction induced by mannitol challenges in participants with asthma on SABA as-needed treatment only was assessed.
  FEV1 baseline was defined as the best FEV1 value (the highest FEV1 of the acceptable efforts) taken pre-mannitol challenge at - 30 min for Visit 2 and Visit 3.
  FEV1 at post-mannitol challenge 2 was the FEV1 result recorded at the end of mannitol challenge 2, i.e. before study intervention treatment, was expected to be at ~490 mins following the mannitol challenge 1.
  If non-inferiority was demonstrated, then comparisons were made to establish the superiority of PT027 versus PT007. The primary efficacy comparison of superiority was based on a 2-sided hypothesis testing approach in the RS. Superiority was concluded if the 2-sided p-value was < 0.05.
Time Frame: Baseline (30 minutes prior to mannitol challenge 1) and at 490 minutes post-mannitol challenge 1
Population: mRS included all participants who were randomized to any of the 2 treatment sequences, A/B or B/A and received any amount of randomized study treatment.
  Treatments A and B were defined as:
  Treatment A = PT027 180/160 μg pMDI Treatment B = PT007 180 μg pMDI
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 16 | 15
milliliters (mL) | 73.4 (317.1) | 137.7 (302.9)

19. Secondary Outcome: Part 2: Peak Fall in FEV1 From Baseline (-30 Min) FEV1 to Post-mannitol Challenge 2, Pre-final Dose of Rescue/Reliever - Non-Inferiority Analysis
Description: as for outcome 17
Time Frame: Baseline (30 minutes prior to mannitol challenge 1) and at 490 minutes post-mannitol challenge 1
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 79 | 79
milliliters (mL) | 246.2 (406.4) | 283.5 (395.8)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in least squares means = -24.52, 95% CI 2-sided [-115.16 to 66.12] — Analysis was performed using linear mixed-effects model. The dependent variable was peak fall in FEV1 derived as FEV1 baseline (- 30 min) - FEV1 result recorded at mannitol challenge 2 completion prior to study intervention (at 490 minutes)

20. Secondary Outcome: Part 2: Peak Fall in FEV1 From Baseline (-30 Min) FEV1 to Post-mannitol Challenge 2, Pre-final Dose of Rescue/Reliever - Superiority Analysis
Description: The protective efficacy of prior repetitive doses of PT027 compared with PT007 on lung function fall in response to a recurring trigger of acute airway obstruction induced by mannitol challenges in participants with asthma on SABA as-needed treatment only was assessed.
  FEV1 baseline was defined as the best FEV1 value (the highest FEV1 of the acceptable efforts) taken pre-mannitol challenge at - 30 min for Visit 2 and Visit 3.
  FEV1 at post-mannitol challenge 2 was the FEV1 result recorded at the end of mannitol challenge 2, i.e. before study intervention treatment, was expected to be at ~490 mins following the mannitol challenge 1.
  If non-inferiority was demonstrated, then comparisons were made to establish the superiority of PT027 versus PT007. The primary efficacy comparison of superiority was based on a 2-sided hypothesis testing approach in the mRS. Superiority was concluded if the 2-sided p-value was < 0.05.
Time Frame: Baseline (30 minutes prior to mannitol challenge 1) and at 490 minutes post-mannitol challenge 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 83 | 85
milliliters (mL) | 246.3 (398.7) | 299.7 (397.1)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Superiority; p = 0.429, Linear mixed effects model; Difference in least squares means = -35.13, 95% CI 2-sided [-123.16 to 52.90] — [estimate comment as in outcome 19, analysis 1]

21. Secondary Outcome: Part 1: Peak Fall in FEV1 From 7 Hours to Post-mannitol Challenge 2, Pre-dose - Non-Inferiority Analysis
Description: The protective efficacy of prior repetitive doses of PT027 compared with PT007 on lung function fall in response to a recurring trigger of acute airway obstruction in participants with asthma on SABA as-needed treatment only was assessed.
  FEV1 baseline was defined as the best FEV1 value (the highest FEV1 of the efforts) taken pre-mannitol challenge at - 30 min for Visit 2 and Visit 3.
  The peak fall in FEV1 (in mL) was derived as: FEV1 at 7 hours (at 420 minutes) post-mannitol challenge 1 - FEV1 result recorded at mannitol challenge 2 completion, before initiation of the study intervention (at 430 minutes).
  The efficacy comparison of non-inferiority of PT027 versus PT007 evaluated the while-on-treatment estimand in the PP analysis set and was based on a 1-sided hypothesis testing approach with a non-inferiority margin of -150 mL.
Time Frame: 420 minutes post-mannitol challenge 1 and 430 minutes post-mannitol challenge 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 15 | 15
milliliters (mL) | 207.5 (222.7) | 272.5 (217.8)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in least squares means = -58.73, 95% CI 2-sided [-139.06 to 21.60] — Analysis was performed using linear mixed-effects model. Dependent variable was peak fall in FEV1 derived as FEV1 7 hours post mannitol challenge1 - FEV1 result recorded at mannitol challenge 2 completion, before initiation of study intervention

22. Secondary Outcome: Part 1: Peak Fall in FEV1 From 7 Hours to Post-mannitol Challenge 2, Pre-dose - Superiority Analysis
Description: The protective efficacy of prior repetitive doses of PT027 compared with PT007 on lung function fall in response to a recurring trigger of acute airway obstruction in participants with asthma on SABA as-needed treatment only was assessed.
  FEV1 baseline was defined as the best FEV1 value (the highest FEV1 of the efforts) taken pre-mannitol challenge at - 30 min for Visit 2 and Visit 3.
  The peak fall in FEV1 (in mL) was derived as: FEV1 at 7 hours (at 420 minutes) post-mannitol challenge 1 FEV1 result recorded at mannitol challenge 2 completion, before initiation of the study intervention (at 430 minutes).
  If non-inferiority was demonstrated, then comparisons were made to establish the superiority of PT027 versus PT007. The primary efficacy comparison of superiority was based on a 2-sided hypothesis testing approach in the RS. Superiority was concluded if the 2-sided p-value was < 0.05.
Time Frame: 420 minutes post-mannitol challenge 1 and 430 minutes post-mannitol challenge 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 16 | 15
milliliters (mL) | 188.9 (227.7) | 272.5 (217.8)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Superiority; p = 0.118, Linear mixed effects model; Difference in least squares means = -61.96, 95% CI 2-sided [-142.16 to 18.24] — [estimate comment as in outcome 21, analysis 1]

23. Secondary Outcome: Part 2: Peak Fall in FEV1 From 480 Minutes to Post-mannitol Challenge 2, Pre-final Dose of Rescue/Reliever - Superiority Analysis
Description: The protective efficacy of prior repetitive doses of PT027 compared with PT007 on lung function fall in response to a recurring trigger of acute airway obstruction in participants with asthma on SABA as-needed treatment only was assessed.
  FEV1 at post-mannitol challenge 2 was the FEV1 result recorded at the end of mannitol challenge 2, i.e. before study intervention treatment, was expected to be at ~490 mins following the mannitol challenge 1.
  If non-inferiority was demonstrated, then comparisons were made to establish the superiority of PT027 versus PT007. The primary efficacy comparison of superiority was based on a 2-sided hypothesis testing approach in the mRS. Superiority was concluded if the 2-sided p-value was < 0.05.
Time Frame: 480 minutes post-mannitol challenge 1 and 490 minutes post-mannitol challenge 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 82 | 85
milliliters (mL) | 425.0 (321.0) | 378.9 (313.4)
Statistical Analysis 1: Comparison: Treatment A (PT027) [Experimental] vs Treatment B (PT007) [Active Comparator]; Statistical Comparison of the Treatment A (PT027) versus Treatment B (PT007); Test type: Superiority; p = 0.241, Linear mixed effects model; Difference in least squares means = 50.39, 95% CI 2-sided [-34.56 to 135.33] — Analysis was performed using linear mixed effects model. Dependent variable was peak fall in FEV1 derived as FEV1 at 480 min - FEV1 result recorded at mannitol challenge 2 completion, before initiation of the study intervention (at 490 min)

24. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The safety and tolerability of repeated dosing of PT027 as compared to PT007 in participants with asthma on SABA as-needed treatment only were assessed.
Time Frame: From Visit 1 until end of follow-up, up to 38 days
Population: Safety analysis set included all participants randomly assigned to any of the 2 study treatment sequences and who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
Number analyzed (Participants) | 100 | 101
Participants
  Any Treatment Emergent Adverse Event (TEAE) | 5 | 4
  Any Treatment Emergent Serious Adverse Event (TESAE) | 0 | 0
  Any TESAE with outcome death | 0 | 0
  Any TEAE leading to discontinuation of IMP | 1 | 0
  Any possibly related TEAE | 2 | 0

ADVERSE EVENTS:
Time Frame: From Visit 1 until end of follow-up, up to 38 days
Description: Safety analysis set included all participants randomly assigned to any of the 2 study treatment sequences and who took at least 1 dose of study treatment.
Arm/Group | Treatment A (PT027) [Experimental] | Treatment B (PT007) [Active Comparator]
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/101
Other Adverse Events (participants affected / at risk) | 5/100 | 4/101
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (PT027) [Experimental] (N=100) | Treatment B (PT007) [Active Comparator] (N=101)
COVID-19 (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information may be disclosed without prior written approval from AstraZeneca

DOCUMENTS (2):
  • Study Protocol (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT05555290/Prot_002.pdf
  • Statistical Analysis Plan (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT05555290/SAP_001.pdf